CLINICAL TRIAL: NCT01328535
Title: Individualized (Timed) Temozolomide Administration as a Means of Immune Reconstitution in Patients With Metastatic Melanoma
Brief Title: Individualized Temozolomide in Treating Patients With Stage IV Melanoma That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1076; NCI-2011-00449 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1076 (Other: Mayo Clinic Cancer Center ID); 10-008497 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2011-03-30; First posted 2011-04-04 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2019-02

CONDITIONS: Recurrent Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — Temozolomide; Flow Cytometry; Coloring Agents; Staining and Labeling; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (individualized chemotherapy) (Experimental): Patients with an established biorhythm receive TMZ PO on recommended day for 5 days. Treatment repeats every 21-42 days until disease progression or unacceptable toxicity. Patients without an established biorhythm receive TMZ PO on days 1-5. Courses repeat every 28 days until disease progression or unacceptable toxicity.
  Interventions: Drug: temozolomide; Other: flow cytometry; Other: staining method; Procedure: biopsy; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: temozolomide — Given PO
  Other Names: SCH 52365; Temodal; Temodar; TMZ
Other: flow cytometry — Correlative studies
Other: staining method — Correlative studies
  Other Names: Staining
Procedure: biopsy — Optional correlative studies
  Other Names: biopsies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This clinical trial studies individualized temozolomide (TMZ) in treating patients with stage IV melanoma that cannot be removed by surgery. Drugs used in chemotherapy, such as TMZ, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving TMZ at different times, which are determined individually for each patient based on the phase (biorhythm) of the immune system response against the tumor may allow for a better drug response and may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To assess the clinical activity of timed administration of TMZ therapy in patients with stage IV melanoma who have or have not received prior chemotherapy for metastatic melanoma. SECONDARY OBJECTIVES: I. To assess the toxicity profile of timed administration of TMZ therapy in patients with stage IV melanoma who have or have not received prior chemotherapy for their metastatic disease. II. To evaluate the parameters of immune homeostasis that are associated with the anti-tumor immune biorhythm in order to gain insight into the mechanism of the observed clinical and immunological effect of timed TMZ chemotherapy. III. To evaluate the impact of timed TMZ chemotherapy on immune biomarkers and the anti-tumor immune biorhythms. OUTLINE: Prior to initiation of therapy patients will undergo a period of immunologic monitoring to analyze the bioperiodicity of their anti-tumor immune response. Patients with an established biorhythm will receive TMZ orally (PO) starting on the recommended day for 5 days. Treatment repeats every 21-42 days (based on the established biorhythm) until of disease progression or unacceptable toxicity. Patients without an established biorhythm are given the option to go off study or receive TMZ PO on days 1-5. Courses repeat every 28 days until disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologic/cytologic proof of stage IV malignant melanoma not amenable to surgery
* Any number of previous chemotherapy regimens (except those containing TMZ or dacarbazine [DTIC]) in the metastatic setting are allowed as long as >= 4 weeks have elapsed from last treatment
* Measurable disease defined as at least one lesion whose longest diameter can be accurately measured as >= 1.0 cm with spiral CT scan, or ≥ 2 cm with computed tomography (CT) component of a positron emission tomography (PET)/CT; Note: disease that is measurable by physical examination only is not eligible
* Life expectancy of >= 3 months
* Eastern Cooperative Oncology Group (ECOG) performance score of 0, 1, or 2
* Recovered from side effects that might interfere with the protocol therapy and: - >= 4 weeks must have elapsed from last radiation treatment to time of study entry - >= 4 weeks must have elapsed from the last chemotherapy administration to time of study entry
* Absolute neutrophil count (ANC) >= 1500/mL
* Platelet count >= 100,000/mcl
* Hemoglobin >= 9gm/mcl
* Creatinine =< 2.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) =< 3 x ULN
* Negative serum pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Ability to understand and the willingness to sign a written informed consent document
* Willingness to return to Mayo Clinic Rochester for follow-up, except for some appointments that can be made with the local physician
* Patient willing to provide research blood samples

Exclusion Criteria:

* Receiving any other investigational agents including those for symptom management
* Uncontrolled intercurrent illness including, but not limited to, the following: - Active infection - Congestive heart-failure (New York Heart Association [NYHA] grade III or IV)
* Pregnant or breast feeding women, or women of child-bearing potential (and/or their partners) who are unwilling to utilize an approved method of birth control during the study and for 1 month afterward
* History of other malignancy < 5 years with the exception of basal cell or squamous cell carcinoma of the skin treated with local resection only, limited stage prostate cancer treated with surgery or radiation therapy with currently undetectable prostate-specific antigen (PSA), or carcinoma in situ of the cervix
* Known standard therapy for the patient's disease that is potentially curative or proven capable of extending life expectancy
* Known immunosuppression (i.e. chronic steroid use) or autoimmune disorder
* Human immunodeficiency virus (HIV) positive
* Current or known history of hepatitis
* Previous treatment with DTIC or TMZ
* Previous immunotherapy treatment for metastatic disease in the preceding 2 months; Note: immunotherapy in the adjuvant setting is allowed
* Previously untreated brain metastases; Note: patients with previously treated brain metastases are allowed as long as these are radiologically stable for >= 3 months and the patient is off steroids for >= 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2013-06-22 (Actual); Study Completion 2018-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roxana Dronca, M.D., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Individualized Chemotherapy)
Started | 25
Completed | 24
Not Completed | 1
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Individualized Chemotherapy)
Number analyzed (Participants) | 24
Age, Continuous [Median (Full Range); unit: years] | 69.5 [36.0 to 84.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival at 4 Months
Description: The distribution of time to progression will be estimated using the method of Kaplan-Meier and the 4 month progression-free rate (percentage) will be provided. Progression is defined as: At least one of the following must be true: At least one new malignant lesion, which also includes any lymph node that was normal at baseline (< 1.0 cm short axis) and increased to ≥ 1.0 cm short axis during follow-up. At least a 20% increase in PBSD (sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes at current evaluation) taking as reference the MSD. In addition, the PBSD must also demonstrate an absolute increase of at least 0.5 cm from the MSD.
Time Frame: Time from registration to the earliest date of documentation of disease progression, assessed at 4 months
Population: Only patients who were evaluable for the primary endpoint were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Treatment (Timed Individualized Chemotherapy): Patients with an established biorhythm receive timed TMZ PO on recommended day for 5 days. Treatment repeats every 21-42 days until disease progression or unacceptable toxicity. Patients without an established biorhythm receive TMZ PO on days 1-5. Courses repeat every 28 days until disease progression or unacceptable toxicity.
Arm/Group | Treatment (Timed Individualized Chemotherapy)
Number analyzed (Participants) | 18
percentage of patients | 22.2 [6.4 to 47.6]

2. Secondary Outcome: Progression-Free Survival
Description: Progression free survival (PFS) is defined as the time from the date of randomization to the date of disease progression or death resulting from any cause, whichever comes first. Progression is defined as:At least one of the following must be true: At least one new malignant lesion, which also includes any lymph node that was normal at baseline (< 1.0 cm short axis) and increased to ≥ 1.0 cm short axis during follow-up. At least a 20% increase in PBSD (sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes at current evaluation) taking as reference the MSD (Section 11.41). In addition, the PBSD must also demonstrate an absolute increase of at least 0.5 cm from the MSD. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Treatment (Untimed Individualized Chemotherapy): Patients with an established biorhythm receive untimed TMZ PO on recommended day for 5 days. Treatment repeats every 21-42 days until disease progression or unacceptable toxicity. Patients without an established biorhythm receive TMZ PO on days 1-5. Courses repeat every 28 days until disease progression or unacceptable toxicity.
Arm/Group | Treatment (Timed Individualized Chemotherapy) | Treatment (Untimed Individualized Chemotherapy)
Number analyzed (Participants) | 18 | 6
months | 3.4 [2.7 to 9.9] | 7.2 [2.5 to NA] — The 95% confidence interval upper bound was not reached.

3. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as the time from randomization to death due to any cause. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Timed Individualized Chemotherapy) | Treatment (Untimed Individualized Chemotherapy)
Number analyzed (Participants) | 18 | 6
months | 23.1 [12.2 to NA] — The 95% confidence interval upper bound was not reached. | 17.5 [12.2 to NA] — The 95% confidence interval upper bound was not reached.

4. Secondary Outcome: Toxicity, Assessed Using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 (v4)
Description: The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns within patient groups. In addition, we will review all adverse event data that is graded as 3, 4, or 5 and classified as either "unrelated" or "unlikely to be related" to study treatment in the event of an actual relationship developing. The overall toxicity rates (percentages) for grade 3 or higher adverse events considered at least possibly related to treatment are reported below.
Time Frame: Up to 2 years
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (Individualized Chemotherapy)
Number analyzed (Participants) | 24
percentage of patients
  Fatigue | 4.2
  Febrile Neutropenia | 8.3
  Neutrophil Count Decreased | 8.3
  Platelet Count Decreased | 25
  Sepsis | 4.2
  Urinary Tract Infection | 4.2
  White Blood Cell Decreased | 8.3
  Abdominal Infection | 4.2

5. Other Pre Specified Outcome: To Evaluate the Impact of Timed TMZ Chemotherapy on Immune Biomarkers and the Anti-tumor Immune Biorhythms.
Time Frame: 6 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: To Evaluate the Parameters of Immune Homeostasis That Are Associated With the Anti-tumor Immune Biorhythm in Order to Gain Insight Into the Mechanism of the Observed Clinical and Immunological Effect of Timed TMZ Chemotherapy
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: The descriptions & grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting. Each CTCAE term in the current version is a unique representation of a specific event used for medical documentation & scientific analysis & is a single MedDRA Lowest Level Term (LLT).
Arm/Group | Treatment (Individualized Chemotherapy)
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 3/24
Other Adverse Events (participants affected / at risk) | 20/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Individualized Chemotherapy) (N=24)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Individualized Chemotherapy) (N=24)
Anemia (Blood and lymphatic system disorders) | 14 (55)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (5)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 5 (6)
Soft tissue infection (Infections and infestations) | 2 (4)
Urinary tract infection (Infections and infestations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 7 (9)
Platelet count decreased (Investigations) | 17 (52)
White blood cell decreased (Investigations) | 8 (10)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (2)
Hypertension (Vascular disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes